CLINICAL TRIAL: NCT02075112
Title: A Pilot Study of Soy Isoflavone, Genistein, in Combination With Radiation Therapy and Cisplatin in Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Soy Isoflavone in Combination With Radiation Therapy and Cisplatin in SCC of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Radiation Therapy Oncology Group (Network)
Responsible Party: Principal Investigator, Kristin Higgins, MD, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00065591; RAD2412-13 (Other: Winship Cancer Institute)
Record Dates: First submitted 2014-02-12; First posted 2014-03-03 (Estimated); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Cancer of Head and Neck
Keywords: Soy; Isoflavone; Radiation Therapy; Cisplatin
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Soybean Proteins; Genistein; Radiation; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Soy isoflavone (Experimental): Study treatment: Soy isoflavone in combination with radiation therapy & cisplatin
  Interventions: Drug: Soy isoflavone; Radiation: Radiation; Drug: Cisplatin

INTERVENTIONS:
Drug: Soy isoflavone — Patients will receive genistein 150 mg daily for the duration of radiation treatment. If a patient is experiencing significant side effects attributable to genistein, the treating physician has the option to reduce genistein to 150 mg every other day.
  Other Names: Genistein
Radiation: Radiation — All patients will undergo computed tomography (CT) simulation with intravenous (IV) contrast unless medical contraindications to IV contrast exist. Gross disease will be treated to 70 Gy in 2 Gy/day.
Drug: Cisplatin — Cisplatin chemotherapy 100 mg/m² on days 1, 22, and 43 of radiation treatment.
  Other Names: Platinol

SUMMARY:
The purpose of this study is to determine if soy supplementation during chemotherapy and radiation therapy will decrease side effects caused by treatment. Long-lasting dry mouth is a side effect of the standard treatment, and we are testing whether soy supplementation during treatment may reduce this symptom and other side effects of chemoradiation.

DETAILED DESCRIPTION:
Concurrent chemoradiation is the standard of care for locally advanced squamous cell carcinoma of the head and neck (SCCHN). Improving the outcome for patients with this disease remains a major challenge.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven squamous cell carcinoma of the head and neck (SCCHN)
* Primary disease site involving the oropharynx
* Clinical stage III or IV
* Age ≥ 18
* Karnofsky Performance Status (KPS) ≥ 70
* Adequate bone marrow, kidney, and hepatic function (no laboratory value > 2 times the normal limit)
* Amylase (0-160 U/L) and lipase (0-130 U/L) levels within 1.5 times the range of normal

Exclusion Criteria:

* Prior history of SCCHN
* Prior history of radiation to the head and neck region
* KPS < 70
* Soy allergy
* Contraindication to cisplatin chemotherapy or plans to alter or reduce cisplatin therapy
* Any head and neck cancer of non-squamous histology
* Any head and neck subsite other than oropharynx (including unknown primary site)
* Patients who are pregnant or lactating
* Patients who may benefit from surgical resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-11; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with grade 2 or higher xerostomia at 1 year post-treatment | 1 year after treatment completion
  The primary outcome of this study is the percentage of patients with symptomatic (grade 2 or higher) xerostomia at 1 year post-treatment, assessed by the Late Effects of Normal Tissues (LENT)/Subjective, Objective, Management, Analytic (SOMA) method.

SECONDARY OUTCOMES:
Exploratory biomarker studies: changes in interleukin 6 | 3 and 6 months post-treatment
  Serum baseline levels of interleukin 6 (IL6) and their levels at 3 and 6 months post-treatment.
Exploratory biomarker studies: changes in vascular endothelial growth factor | 3 and 6 months post-treatment
  Serum baseline levels of vascular endothelial growth factor (VEGF) and their levels at 3 and 6 months post-treatment.
Exploratory biomarker studies: changes in isoprostanes levels | 3 and 6 months post-treatment
  Baseline urinary levels of isoprostanes before treatment, and 3 and 6 months post-treatment, as a potential marker of oxidative stress associated with chemoradiation.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Higgins, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia